CLINICAL TRIAL: NCT00068471
Title: Phase I-II Study of the Safety, Tolerance and Pharmacokinetics of Anidulafungin in Immunocompromised Children With Neutropenia
Brief Title: Anidulafungin in Treating Immunocompromised Children With Neutropenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000322888; NCI-03-C-0229C; NCT00063466 (obsolete NCT alias)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-04

CONDITIONS: Infection; Neutropenia; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: infection; neutropenia; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Infections; Neutropenia | interventions — Anidulafungin

INTERVENTIONS:
Drug: anidulafungin

SUMMARY:
RATIONALE: Anidulafungin may be effective in preventing fungal infections in immunocompromised children who have neutropenia.

PURPOSE: This phase I/II trial is studying the side effects of anidulafungin and to see how well it works in preventing fungal infections in immunocompromised children with neutropenia caused by chemotherapy or aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety, tolerability, and pharmacokinetics of anidulafungin in immunocompromised children with neutropenia.
* Determine the frequency of deeply invasive fungal infections in children receiving this drug for early empirical therapy.

OUTLINE: This is a dose-escalation, open-label, multicenter study. Patients are assigned to 1 of 2 groups according to age (2 to 11 years vs 12 to 17 years).

Patients receive anidulafungin IV once daily over 45-120 minutes. In both groups, cohorts of 6 patients receive escalating doses of anidulafungin. Treatment continues for up to 28 days or until patients recover from neutropenia or become eligible for standard empirical antifungal therapy in the absence of unacceptable toxicity or breakthrough fungal infection.

Patients are followed at 7-9 days.

PROJECTED ACCRUAL: A total of 25 patients (approximately 12 per group) were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Neutropenia due to cytotoxic chemotherapy or aplastic anemia

  * Duration expected to be 10 days
  * Absolute neutrophil count less than 500/mm^3 OR less than 1,000/mm^3 and expected to fall below 500/mm^3 within 72 hours
* No deeply invasive fungal infection confirmed prior to study entry

PATIENT CHARACTERISTICS:

Age

* 2 to 17

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* AST or ALT no greater than 5 times upper limit of normal (ULN)
* Bilirubin no greater than 2.5 times ULN

Renal

* Creatinine clearance at least 30 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 30 days after study participation
* No prior anaphylaxis attributed to the echinocandin class of antifungals
* No other concurrent medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 4 weeks since prior investigational drugs
* No prior participation in this clinical trial
* No prior anidulafungin
* No other concurrent investigational drugs
* No other concurrent systemic antifungal agents (e.g., amphotericin, systemic azoles, or triazole antifungal agents)

  * Concurrent oral, nonabsorbable azoles and topical antifungal agents (e.g., nystatin and/or azole formulations) allowed
* Concurrent broad-spectrum antibiotics allowed

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-07; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Walsh, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee